CLINICAL TRIAL: NCT00655915
Title: Corticosteroid Injection as a Predictor of Outcome in Carpal Tunnel Release
Status: Terminated | Type: Observational
Why Stopped: Study was terminated by principal investigator
Sponsor: Vanderbilt University (Other)
Responsible Party: Jeffry T. Watson, MD / Assistant Professor of Orthopaedic Surgery, Vanderbilt University Medical Center
Other Study IDs: 071107
Record Dates: First submitted 2008-03-28; First posted 2008-04-10 (Estimated); Last update posted 2011-03-09 (Estimated); Status verified 2011-03

CONDITIONS: Carpal Tunnel Syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Adrenal Cortex Hormones; Betamethasone; Lidocaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Injection Patients: Those patients who receive corticosteroid injections for carpal tunnel syndrome
  Interventions: Other: Corticosteroid Injection- 1ml of Betamethasone and 1 ml of 1% Lidocaine

INTERVENTIONS:
Other: Corticosteroid Injection- 1ml of Betamethasone and 1 ml of 1% Lidocaine — Patients will receive a carpal tunnel injection of 1 mg of betamethasone and 1 mL of 1% lidocaine will be infiltrated by small gauge (ie. 25- or 27-gauge) needle via attending surgeon preference. These are routinely performed by injecting 1cm proximal to distal wrist crease just ulnar to palmaris longus tendon although multiple techniques have been described. Elicitation of median nerve symptoms during needle placement requires redirecting needle prior to injection to avoid median nerve infiltration.

SUMMARY:
This study will investigate whether symptomatic improvement following carpal tunnel corticosteroid injection can be correlated to symptomatic improvement following carpal tunnel release and therefore serve as a prognostic indicator.

Clinical question: Does response to corticosteroid injection in CTS predict outcomes of surgical treatment?

Secondary Questions:

1. Can we confirm previous retrospectively collected data that a certain percentage of conservatively managed patients with steroid injection will avoid surgery, and that patients who undergo surgery will have better outcomes than those who do not.
2. Are there differences between worker's compensation and non-worker's compensation patients with regard to the primary clinical question?
3. What are Carpal Tunnel Release outcomes for the subset of patients with negative electrophysiologic studies?
4. What are the outcomes of patients who undergo carpal tunnel release vs. those who choose not to undergo carpal tunnel release?

A prospective cohort design study is the appropriate study design in order to measure the association between a predictor (response to injection) and outcome (response to surgery).

DETAILED DESCRIPTION:
Carpal Tunnel Syndrome is a painful condition that is caused by compression of the median nerve in the wrist. Symptoms usually are pain, weakness, or numbness in the hand and wrist, radiating up the arm. Corticosteroid injections have been utilized in the conservative management of carpal tunnel syndrome for several decades. They have been shown to be relatively safe with a very low reported complication rate. Recent efforts in the literature have shown they are efficacious for a majority of patients although their effects are usually transient. Several studies have attempted to show a predictive value of corticosteroid injection with regard to who will ultimately benefit from carpal tunnel release. There is a trend towards positive predictability with several retrospective studies showing that patients who have a clinical benefit from steroid injection are more likely to have a successful outcome from carpal tunnel release. Carpal tunnel release remains the definitive treatment option for carpal tunnel syndrome, and a clinical test which could give the practitioner and patient additional information regarding likelihood of successful outcome of surgery would be a valuable prognostic tool.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a clinical diagnosis of carpal tunnel syndrome
* English speaking patients only

Exclusion Criteria:

* Patients less than 18 years old
* Patients who are pregnant by patient report or intending to become pregnant during the study
* Patients unwilling or unable to return for follow-up visits prescribed by the study protocol.
* Patients who qualify for inclusion in the study, but refuse to participate.
* Patients with evidence of thenar atrophy on exam
* Patients with a diagnosis of peripheral neuropathy or other neuropathy.
* Patients with previous ipsilateral carpal tunnel injection or release.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who present to Vanderbilt Hand Center with carpal tunnel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-12; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffry T Watson, M.D., Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt Hand & Upper Extremity Center, Nashville, Tennessee, United States